CLINICAL TRIAL: NCT01706354
Title: Does Regional Compared to Local Anaesthesia Influence Outcome After Arteriovenous Fistula Creation?
Brief Title: Local Anaesthesia vs Regional Block for Arteriovenous Fistulae
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Emma Aitken (Other)
Collaborators: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor-Investigator, Emma Aitken, Clinical Research Fellow Department of Renal Surgery, NHS Greater Glasgow and Clyde
Organization: NHS Greater Glasgow and Clyde (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 12/WS/0199
Record Dates: First submitted 2012-10-03; First posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-10

CONDITIONS: End Stage Renal Disease
Keywords: end stage renal disease; vascular access; regional anaesthesia
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local anaesthetic (Active Comparator): Infiltration of local anaesthetic into the surgical site by the surgeon using a combination of 0.5% L-bupivicaine prior to incision and 1% lignocaine topically after the wound is opened. Maximum dose limits of 2mg/kg for bupivicaine, and 3mg/kg for lignocaine will be observed, recognising that these are additive.
  Interventions: Procedure: Local Anaesthetic
- Regional anaesthetic (Experimental): Ultrasound guided brachial plexus block. Supraclavicular will be the block performed unless there is a contraindication in which case axillary block may be used. A 1:1 mixture of 0.5% L-bupivicaine and 1.5% lignocaine with adrenaline (1 in 200,000) will be injected, up to a volume of 40ml but using a minimum of 25ml. Maximum dose limits of 2mg for bupivicaine and 7mg/kg for lignocaine with adrenaline will be observed, recognising that these are additive.
  Interventions: Procedure: Regional anaesthetic

INTERVENTIONS:
Procedure: Local Anaesthetic — Infiltration of local anaesthetic into the surgical site by the surgeon using a combination of 0.5% L-bupivicaine prior to incision and 1% lignocaine topically after the wound is opened. Maximum dose limits of 2mg/kg for bupivicaine, and 3mg/kg for lignocaine will be observed, recognising that these are additive.
  Arms: Local anaesthetic
Procedure: Regional anaesthetic — Ultrasound guided brachial plexus block. Supraclavicular will be the block performed unless there is a contraindication in which case axillary block may be used. A 1:1 mixture of 0.5% L-bupivicaine and 1.5% lignocaine with adrenaline (1 in 200,000) will be injected, up to a volume of 40ml but using a minimum of 25ml. Maximum dose limits of 2mg for bupivicaine and 7mg/kg for lignocaine with adrenaline will be observed, recognising that these are additive.
  Arms: Regional anaesthetic

SUMMARY:
End stage renal failure (ESRF)describes an irreversible loss in renal function. The majority of these patients will opt for haemodialysis (HD)as their chosen method of renal replacement therapy (RRT). Arteriovenous fistulae (AVF) are the optimal method of achieving vascular access to permit HD. AVF are created with a small surgical procdure to join the artery and vein together. Over the next 6- 8weeks after surgery the AVF should grow ("mature") into a vessel suitable for needles to be inserted for dialysis. Unfortunately however, around 24% - 35% of AVF fail at an early stage. Some anaesthetic techniques can influence intraoperative blood flow and venous diameter, factors which are associated with fistula success. There remains no conclusive evidence that any particular anaesthetic technique can significantly influence long term surgical outcome. This study aims to investigate whether a regional, compared to local, anaesthetic technique can affect fistula patency.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) describes abnormal kidney structure or function and is a significant public health problem. It is common, increasingly prevalent with age and often co-exists with significant morbidities, such as diabetes mellitus, hypertension, hyperlipidaemia, cerebrovascular disease and coronary artery disease. Patients with a diagnosis of CKD have a decreased life expectancy compared with individuals without this diagnosis. This is primarily due to cardiovascular disease, but other complications of CKD include bone and mineral disorders, anaemia, depression, and malnutrition. Early recognition and treatment of these complications is recommended.

In a proportion of patients, CKD will progress to end stage renal disease (ESRD). This is defined as an irreversible decline in kidney function for which renal replacement therapy (RRT) is required if the patient is to survive. In one UK study, 4% of patients with CKD progressed to develop ESRD requiring RRT over a five and a half year follow up period. The decision to commence RRT takes into account symptoms of biochemical disturbance, in conjunction with the risks and inconvenience of starting RRT. European Best Practice Guidelines recommend that RRT should commence when the estimated Glomerular Filtration Rate (eGFR) falls below 15ml/min/1.73m2 or when symptoms of uraemia, fluid overload or malnutrition are resistant to medical therapy. In an asymptomatic patient, an eGFR of below 6ml/min/1.73m2 would also prompt the initiation of dialysis. It is known that the life expectancy of patients receiving RRT is shorter than that of the general population and varies further dependent on underlying diagnosis and age. For example, the median survival for a patient in Scotland aged 45 - 64 years starting RRT for glomerulonephritis is 7.7 years, whereas the median survival of a patient in the same age group with a diagnosis of diabetic nephropathy is 2.9 years. The life expectancy of a male of the same age group within the general Scottish population is 24.2 years. Instituting RRT prolongs life and reduces the incidence of vasculo-occlusive events in patients with ESRD. As such, patients with CKD should be monitored by a nephrologist in order that timely referral for preparation for RRT can be made.

Renal replacement therapy may come in the form of haemodialysis, peritoneal dialysis or renal transplantation, and may be managed both in and out of hospital. Haemodialysis (HD) remains the most common modality of first RRT in Scotland; of 2885 patients commencing RRT during the period 2005-2009, 2264 received HD. In order to undergo HD, there must be a connection between the patient's vascular system and the dialysis machine. The most common method is surgical creation of an arteriovenous fistula (AVF), into which a needle can be inserted that in turn is connected to a dialysis machine. In 2009, 75% of Scottish patients undergoing HD underwent formation of an arteriovenous fistula (AVF). Other options for vascular access include arteriovenous grafts using synthetic materials and long-term central venous catheters, though these are associated with higher rates of occlusive and infective complications. AVF are currently regarded as the optimal form of vascular access for HD and are recommended by National guidelines. There is excellent evidence that good quality, stable vascular access is a major factor in determining survival in this group of CKD patients. Unfortunately however, around 24% - 35% of arteriovenous fistulae (AVF) fail at an early stage. Some anaesthetic techniques can influence intraoperative blood flow and venous diameter, factors which are associated with fistula success. There remains no conclusive evidence that any particular anaesthetic technique can significantly influence long term surgical outcome. This study aims to investigate whether a regional, compared to local, anaesthetic technique can affect fistula patency.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Adult patients >18 years old
* Competent to give consent
* Scheduled for primary AVF formation at either radial or brachial artery.

Exclusion Criteria:

* Allergy to local anaesthetic.
* Coagulopathy
* Infection at the anaesthetic or surgical site.
* Patient preference for general or alternative anaesthesia
* Significant peripheral neuropathy or neurologic disorder affecting the upper extremity
* Pregnancy
* Previous AVF creation
* Known cephalic vein occlusion, central vein stenosis, brachial or radial artery stenosis
* Vein or artery less than 1.8mm, as measured by ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Primary patency | 3 months
  Primary patency defined as unequivocal maturation to permit cannulation with thrill and bruit without intervention (Y/N)

SECONDARY OUTCOMES:
Immediate Patency | 1 hours post-operatively
  Defined as the unequivocal presence of thrill and bruit in the fistula in recovery room 1 hour post-opertaively (Y/N)
Primary patency | 1 month, 1year
  Defined as the unequivoval presence of a thrill/ bruit at 1 month/ 1 year (Y/N)
Functional patency | 1, 3 and 12 months
  Defined as a fistula capable of sustaining two needles haemodialysis for at least 6 consecutive sessions without intervention(Y/N)
Secondary patency | 3 and 12 months
  Defined as a fistula suitable to sustain haemodialysis only after additional intervention (e.g. revisional surgery/ angioplasty)
Ultrasound flows in brachial artery | Pre-/post anaesthetic, 1, 3 and 12 months
Patient satisfaction | 24 hours
Success of anaesthetic | Immediate
  Complications and efficacy (VAS for pain)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Clancy, MBBS FRCS, Principal Investigator — NHS Greater Glasgow and Clyde
Locations (1):
- Department of Renal Surgery, Western Infirmary, Glasgow, United Kingdom

REFERENCES:
- [Derived] Aitken E, Kearns R, Gaianu L, Jackson A, Steven M, Kinsella J, Clancy M, Macfarlane A. Long-Term Functional Patency and Cost-Effectiveness of Arteriovenous Fistula Creation under Regional Anesthesia: a Randomized Controlled Trial. J Am Soc Nephrol. 2020 Aug;31(8):1871-1882. doi: 10.1681/ASN.2019111209. Epub 2020 Jul 24. PMID 32709710
- [Derived] Aitken E, Jackson A, Kearns R, Steven M, Kinsella J, Clancy M, Macfarlane A. Effect of regional versus local anaesthesia on outcome after arteriovenous fistula creation: a randomised controlled trial. Lancet. 2016 Sep 10;388(10049):1067-1074. doi: 10.1016/S0140-6736(16)30948-5. Epub 2016 Aug 1. PMID 27492881
- [Derived] Macfarlane AJ, Kearns RJ, Aitken E, Kinsella J, Clancy MJ. Does regional compared to local anaesthesia influence outcome after arteriovenous fistula creation? Trials. 2013 Aug 19;14:263. doi: 10.1186/1745-6215-14-263. PMID 23958289